CLINICAL TRIAL: NCT03111004
Title: BeyondSilos - Integrated Care Leading to a More Personalised and Coordinated Care, Improving Outcomes for Elderly Patients, Delivering More Effective Care and Support, and Provide More Cost Efficient Health and Social Services
Brief Title: BeyondSilos - More Personalised and Coordinated Care and Improved Outcomes for Elderly Patients
Acronym: BeyondSilos
Status: Completed | Type: Observational
Sponsor: Him SA (Other)
Responsible Party: Sponsor
Other Study IDs: BeyondSilos_CIP_No.621069
Record Dates: First submitted 2017-03-07; First posted 2017-04-12 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Heart Failure; Stroke; COPD; Diabetes
Keywords: information technology; telemedicine; integrated care; MAST framework; organizational change; social care; elderly patients
MeSH Terms: conditions — Heart Failure; Stroke; Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The Study Group receives 'new care' (integrated health and social care)
  Interventions: Other: New Care
- Comparator Group: The comparator group receives usual care

INTERVENTIONS:
Other: New Care — All settings that are in any way relevant to the provision of health and social care are integrated, including: out-of-hospital (community) services as well as hospitals, GPs' offices, community nurses, and any type of care practitioners, users' homes and volunteer service providers' offices
  Other Names: integrated health care and social care
  Groups: Study Group

SUMMARY:
The study evaluates the impact of the new organisational models developed in the framework of the BeyondSilos pilot service in order to provide ICT supported integrated health and social care to elderly patients

DETAILED DESCRIPTION:
The overall aim of the evaluation carried out in BeyondSilos is to identify the differences introduced by implementing ICT supported integrated care in different domains according to the MAST evaluation framework, including safety, clinical and social outcomes, resource use and cost of care, user/carer experience and organisational changes.

The focus of the evaluation will be the impact of so called "horizontal" integration, which is the integration between social care and health care, and the changing organisational models for elderly patients.

The hypothesis in this study is that integrated care (IC) will lead to a more personalised and coordinated care, improve outcomes for elderly patients, deliver more effective care and support, and provide more cost efficient health and social services.

ELIGIBILITY:
Potential participants are selected by screening electronic healthcare and social care records or/and the hospital / national databases and/or during long term condition annual reviews in the community setting. If necessary, candidates are informed about the nature and the objectives of the evaluation. If a candidate passes the inclusion/exclusion criteria and signs the informed consent form, if necessary, they participate in the evaluation.

Inclusion Criteria:

* Age ≥65 years.
* Presence of health needs specified as: Presence of heart failure, stroke, COPD or diabetes (diagnosed at hospital or at specialist visit) plus at least one additional chronic disease / condition included in the Charlson Comorbidity Index (CCI).
* Presence of social needs based on Barthel Index of Activities of Daily Living and Instrumental Activities of Daily Living (IADL).
* Reasonable expectation of permanence in the BeyondSilos project for the whole data collection period (18 months).
* Informed consent, signed if necessary (by the subject or his/her delegate).
* Capability to handle ICT equipment / devices alone, or with the help from a delegate.
* Presence of good/reliable communication connection at home (internet, telephone or what is needed for the ICT connection).

Exclusion Criteria:

Subjects who have been registered with an active cancer diagnosis and undergoing treatment, has undergone an organ transplant, or is undergoing dialysis prior to enrolment.

* Subjects in a terminal state
* People with an AIDS diagnose.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly living independently at home with diagnosed chronic disease(s).
Sampling Method: Probability Sample
Enrollment: 1840 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Change in length of the hospital stay | Days between admission and discharge of patient's admission episodes, measured based on follow up during whole length of study and accumulated at END of study (at month 18)
  Change in the duration of hospitalization (calculated from admission date and discharge date) measured in days

SECONDARY OUTCOMES:
Re-hospitalisation period | Days between last discharge of patient and her/his re-hospitalization, measured based on follow up during whole length of study and accumulated at END of study (at month 18)
  Re-hospitalisation within 30 days (calculate from admission date and discharge date) measured in days
Patient encounters | Number of registered encounters/contacts between patient and GP, Specialists, Nurse, other involved healthcare providers within the timeframe based on total count in period between start (month 0) end (month 18) of study
  Encounters and contacts between patient and GP, Specialists, Nurse, other involved healthcare providers
Weight | Weight measured in kilo grams (kg) at baseline (month 0) and at end (month 18) of study duration
  Weight as disease specific health status measurement
Blood pressure | Blood pressure measured in mmHg at baseline (month 0) and at end (month 18) of study duration
  Blood pressure as disease specific health status measurement
Heart rate | Heart rate measured in beats per minute (bpm) at baseline and at end of study duration
  Heart rate pressure as disease specific health status measurement
Oxygen saturation | Oxygen saturation measured in SpO2 (or %) based on measurement at baseline (month 0) and at end (month 18) of study duration
  Oxygen saturation pressure as disease specific health status measurement
Blood glucose | Blood glucose measured in mg/dl based on measurement at baseline (month 0) and at end (month 18) of study duration
  Blood glucose pressure as disease specific health status measurement
HbA1c | HbA1c measured in percentage (%) based on measurement at baseline and at end of study duration
  HbA1c pressure as disease specific health status measurement
Creatinine | Creatinine measured in mg/dl based on measurement at baseline (month 0) and at end (month 18) of study duration
  Creatinine pressure as disease specific health status measurement
Charlson Comorbidity Index (CCI) | Charlson Comorbidity Index (CCI) measured in (a) ICD-10-CM and (b) CCI scale based on measurement at baseline (month 0) and at end (month 18) of study duration
  Charlson Comorbidity Index (CCI) as a generic health related / functional quality of life
Barthel index | Barthel index measured in index scale based on measurement at baseline (month 0) and at end (month 18) of study duration
  Barthel index as a generic health related / functional quality of life
Self-maintaining and instrumental activities of daily living (IADL) | Self-maintaining and instrumental activities of daily living (IADL) measured in (IADL) scale based on measurement at baseline (month 0) and at end (month 18) of study duration
  Self-maintaining and instrumental activities of daily living (IADL) as a generic health related / functional quality of life
Geriatric Depression Scale (GDS Short Form) | GDS measured in GDSsf-scale based on measurement at baseline (month 0) and at end (month 18) of study duration
  Geriatric Depression Scale (GDS Short Form) as a psychological measure
Anxiety and depression based on HADS | Anxiety and depression according to HADS-scale measurements based on measurement at baseline (month 0) and at end (month 18) of study duration
  Anxiety and depression (according to HADScale) as a psychological measure
PIRU questionnaire on user experience (selected questions) of Integrated Care (IC) | User experience (PIRU) measurements based on PIRU-scale measurement at baseline and at end of study duration
  PIRU questionnaire on user experience of IC as a user perspectives measure
End user perception of service utility according to eCCIS (selected questions) | End user perception of service utility based on eCCIS-scale measurement at baseline (month 0) and at end (month 18) of study duration
  End user perception of service utility (eCCIS) as a user perspectives measure
Carer perception of service utility according to eCCIS (selected questions) | Carer perception of service utility based on eCCIS-scale measurement at baseline (month 0) and at end (month 18) of study duration
  Carer perception of service utility (eCCIS) as a user perspectives measure

CONTACTS AND LOCATIONS:
Overall Officials: Panos A Stafylas, Study Director — Him SA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vandenbroucke JP, von Elm E, Altman DG, Gotzsche PC, Mulrow CD, Pocock SJ, Poole C, Schlesselman JJ, Egger M; STROBE Initiative. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): explanation and elaboration. Int J Surg. 2014 Dec;12(12):1500-24. doi: 10.1016/j.ijsu.2014.07.014. Epub 2014 Jul 18. PMID 25046751
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Background] Berger ML, Dreyer N, Anderson F, Towse A, Sedrakyan A, Normand SL. Prospective observational studies to assess comparative effectiveness: the ISPOR good research practices task force report. Value Health. 2012 Mar-Apr;15(2):217-30. doi: 10.1016/j.jval.2011.12.010. PMID 22433752
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Derived] Piera-Jimenez J, Daugbjerg S, Stafylas P, Meyer I, Muller S, Lewis L, da Col P, Folkvord F, Lupianez-Villanueva F. BeyondSilos, a Telehealth-Enhanced Integrated Care Model in the Domiciliary Setting for Older Patients: Observational Prospective Cohort Study for Effectiveness and Cost-Effectiveness Assessments. JMIR Med Inform. 2020 Oct 6;8(10):e20938. doi: 10.2196/20938. PMID 33021490
- See also: Project Website BeyondSilos — http://beyondsilos.eu/project/